CLINICAL TRIAL: NCT06009107
Title: A Phase I/II, Single Arm, Multi-center Study Evaluating the Safety and Efficacy of HY004 in Adult Patients With Relapsed/Refractory B-precursor Acute Lymphoblastic Leukemia (r/r B-ALL)
Brief Title: A Study of HY004 Treatment in Adult Relapsed/Refractory B-precursor Acute Lymphoblastic Leukemia (r/r B-ALL)
Acronym: B-ALL
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor changed product development plan
Sponsor: Juventas Cell Therapy Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HY004101
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
Keywords: HY004; Cluster of differentiation antigen 19 and/or 22(CD19 and/or 22); CD19/22-directed CAR-T cells
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Cyclophosphamide; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant Group (Experimental): Participants with relapsed or refractory B-precursor acute lymphoblastic leukemia (r/r B-ALL) will receive conditioning chemotherapy (fludarabine 25-30 mg/m^2 intravenously [IV] over 30 minutes on Day -5, Day -4, and Day -3 and cyclophosphamide 500 mg/m^2 IV over 60 minutes on Day -5, Day -4), following a single IV infusion of chimeric antigen receptor (CAR) transduced autologous T cells(HY004).
  Interventions: Biological: HY004; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate

INTERVENTIONS:
Biological: HY004 — A single infusion of Autologous 2nd generation CD19/CD22-directed CAR-T cells administered intravenously.
Drug: Cyclophosphamide — Administered intravenously.
Drug: Fludarabine Phosphate — Administered intravenously.

SUMMARY:
This is a multi-center, phase I/II trial to evaluate the safety and efficacy of HY004 treatment in Adult patients with relapsed or refractory B-cell acute lymphoblastic leukemia (r/r B-cell ALL).

DETAILED DESCRIPTION:
This trial is a multi-center, open label, single-arm, phase I/II trial to evaluate the safety and efficacy of HY004 treatment in Adult (aged 18~65 years old) patients with r/r B-cell ALL.

The phase I part of the trial is to evaluate the safety, optimal dose of HY004, Pharmacokinetics/Pharmacodynamics(PK/PD)and preliminary efficacy in the treatment of Adult patients with r/r B-cell ALL. The phase II part of the trial is to evaluate the efficacy and safety of HY004 in in the treatment of Adult patients with r/r B-cell ALL. The study includes screening, pre-treatment (Cell Product manufacture & lymphodepletion), HY004 infusion, safety and efficacy follow-up, and survival follow-up. All subjects who have received HY004 infusion will be followed for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent prior to any study procedures (patient and/or parent or legal guardian);
2. Gender is not limited, and the age at the time of screening is ≥ 18 years old and ≤ 65 years old;
3. Relapsed or refractory acute lymphoblastic leukemia (ALL);
4. Documentation of CD19 and/orCD22 tumor expression demonstrated in bone marrow or peripheral blood within 3 months before screening;
5. Bone marrow with ≥ 5% lymphoblasts by morphologic assessment at screening;
6. ECOG score 0-1 points;
7. Organ function requirements: All patients must have adequate renal and liver functions.

Exclusion Criteria:

1. Active Central Nervous System (CNS) involvement by malignancy;
2. Isolated extra-medullary disease relapse;
3. Patients with Burkitt's lymphoma/leukemia;
4. History of concomitant genetic syndrome;
5. Patients with acute graft-versus-host disease (GVHD) or moderate-tosevere chronic GVHD within 4 weeks before screening; Patients with a history of allogeneic hematopoietic stem cell transplantation within 12 weeks before single collection;
6. Active systemic autoimmune disease;
7. Known infection with human immunodeficiency virus (HIV) or chronic infection with hepatitis B virus (HbsAg positive) or hepatitis C virus (anti- HCV positive);
8. Patients with active infections at screening;
9. Patients who have used CAR-T cell therapy before screening;
10. Patients with an expected lifespan of less than 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall Remission Rate (ORR) | at the end of Month 3
  ORR is defined as Complete Remission (CR) and Complete Remission with Incomplete Blood Count Recovery (CRi) per NCCN classification, as determined by Independent Review Committee (IRC).

SECONDARY OUTCOMES:
Overall Remission Rate (ORR) | within 3 months
  ORR is defined as Complete Remission (CR) and Complete Remission with Incomplete Blood Count Recovery (CRi) per NCCN classification.
Best overall response (BOR) | up to 2 years
  The proportion of patients who have achieved the best response (CR or CRi) after HY004 treatment.
Overall Remission Rate (ORR) with minimal residual disease (MRD) negativity | at the end of Month 3
  Overall Remission Rate (ORR) with minimal residual disease (MRD) negativity as determined by IRC and Investigators; MRD negativity as determined using flow cytometry.
Duration of remission (DOR) | to data cutoff date
  DOR is defined as the time between their first complete response per independent review to relapse or any death in the absence of documented relapse.
Allogeneic Stem Cell Transplant (Allo-SCT) rate | First infusion date of HY004 to data cutoff date(up to 2 years)
  The proportion of patients who have received Allo-SCT after HY004 treatment.
Relapse Free Survival (RFS) | up to 2 years
  RFS is defined as the time from the HY004 infusion date to the date of disease relapse or death from any cause.
Event-Free Survival(EFS) | up to 2 years
  EFS is defined as the time from the HY004 infusion date to the date of any event, including disease progression, cessation of treatment for any reason, or death.
Overall survival (OS) | 2 years
  OS is defined as the time from the HY004 Cell Injection infusion to the date of death from any cause.
Percentage of Participants Experiencing Treatment-Emergent Adverse Events（TEAE） | up to 2 years
  Evaluate the type, frequency, severity of adverse events, and abnormal laboratory test values; Evaluate the frequency and severity of adverse events related to HY004.

OTHER OUTCOMES:
In vivo cellular Pharmacokinetic (PK) profile of HY004 in units of transgene copy number per genomic DNA (gDNA) amount. | Up to 3 months(BM sample); Up to 2 years(Blood sample)
  To characterize the in vivo cellular pharmacokinetic (PK) profile (levels, persistence, trafficking) of HY004 cells in target tissues (blood, bone marrow andCerebral Spinal Fluid (CSF)if available)by quantitative polymerase chain reaction(qPCR).
In vivo cellular Pharmacokinetic (PK) profile of HY004 in units of percent of CAR-positive cells. | Up to 3 months(BM sample); Up to 2 years(Blood sample)
  To characterize the in vivo cellular pharmacokinetic (PK) profile (levels, persistence, trafficking) of HY004 cells in target tissues (blood, bone marrow andCerebral Spinal Fluid (CSF)if available)by Flow Cytometry.
In vivo cellular pharmacodynamics (PD) profile of HY004. | 28 days
  To characterize the concentration of cytokines ,including Interleukin-6(IL-6) at least in Serum.
Prevalence and incidence of humoral immunogenicity to HY004. | 2 years
  To characterize the concentration of anti-drug antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang M.D., Principal Investigator — Study Principal Investigator Institute of Hematology & Blood Diseases Hospital

IPD SHARING:
Plan to Share IPD: No
Currently the investigators have no plan of interim anaylsis, the investigators don't plan to share individual participant data(IPD) during the trial on-going.